CLINICAL TRIAL: NCT04806607
Title: 19Gauge Fine Needle Biopsy (FNB) Versus 22Gauge FNB for Endoscopic Ultrasound Guided Liver Biopsy (EUS-LB): A Randomized Prospective Trial
Brief Title: 19Gauge Fine Needle Biopsy (FNB) Versus 22Gauge FNB for Endoscopic Ultrasound Guided Liver Biopsy (EUS-LB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, David L. Diehl, Principal Investigator, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1072
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized trial comparing the biopsy specimen adequacy of 19G versus 22G core needles in subjects undergoing an EUS-LB.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 19Gauge Fine Needle Biopsy (Active Comparator): 19Gauge Fine Needle
  Interventions: Procedure: 19G FNB; Procedure: 22G FNB
- 22 Gauge Fine Needle Biopsy (Active Comparator): 22Gauge Fine Needle
  Interventions: Procedure: 19G FNB; Procedure: 22G FNB

INTERVENTIONS:
Procedure: 19G FNB — Biopsy specimen adequacy using the 19G FNB
Procedure: 22G FNB — Biopsy specimen adequacy using the 22G FNB.

SUMMARY:
To determine the adequacy of EUS-LB using a 19G core needle compared to a 22G core needle in a prospective randomized study.

DETAILED DESCRIPTION:
The 19Gauge core and 22Gauge core needles have both been used for EUS-LB with good success. Previous studies have reported good safety and tissue adequacy with both the needles, but the head-on comparison between these two needles is lacking.

This is a prospective randomized trial comparing the biopsy specimen adequacy of 19Gauge versus 22Gauge core needles for EUS-LB.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing EUS-LB
* Platelet Count > 50,000
* International normalized ratio (INR) < 1.5
* Age > 18 years of age
* Non-Pregnant Patients

Exclusion Criteria:

* Age < 18 Years of Age
* Pregnant Patients
* Inability to obtain consent
* Anticoagulants or anti-platelet agents (excluding aspirin) within the last 7 -10 days
* Platelet count < 50,000
* Presence of Ascites
* Known Liver Cirrhosis

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Length of Longest Piece | Up to 5 Days
  Length of the longest piece of the liver tissue obtained

SECONDARY OUTCOMES:
Aggregate Specimen Length | 3 to 5 Days
  Cumulative length of all the pieces of tissue obtained
Degree of Fragmentation | 3 to 5 Days
  Size of the fragments of the samples will be measured, then classified as small (<5 mm), medium (5-8 mm) or large (>8 mm), then compared for the 2 needles
Number of Portal Tracts in the Specimen | 3 to 5 Days
  Number of portal triads will be counted in the specimens and compared for the 2 needles
Adverse Events and Serious Adverse Events | 7 to 10 Days Post Procedure
  Untoward, undesired, or unplanned event

CONTACTS AND LOCATIONS:
Overall Officials: David L Diehl, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diehl DL, Sangwan V, Johal AS, Khara HS, Confer B. Comparing a 19-gauge fine-needle biopsy needle with a 22-gauge fine-needle biopsy needle for EUS-guided liver biopsy sampling: a prospective randomized study. Gastrointest Endosc. 2024 Jun;99(6):931-937. doi: 10.1016/j.gie.2023.12.022. Epub 2023 Dec 21. PMID 38141686